CLINICAL TRIAL: NCT03541499
Title: A Phase 2A Partially-Blind Placebo Controlled Trial to Evaluate the Safety and Immunogenicity of Live Attenuated, Intranasal B. Pertussis Vaccine (BPZE1) in Healthy Adults
Brief Title: Safety and Immunogenicity of Intranasal BPZE1 Vaccination in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17-0010
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Results first posted 2022-02-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2021-08-18

CONDITIONS: Pertussis; Pertussis Immunisation
Keywords: B. pertussis Vaccine; BPZE1; Immunogenicity; Safety
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Experimental): 800 microliters (10^7 CFU) of B. pertussis vaccine (BPZE1) administered intranasally with the VaxINator device on Day 1, n=15
  Interventions: Biological: BPZE1
- Group 2 (Experimental): 800 microliters (10^9 CFU) of BPZE1 administered intranasally with the VaxINator device on Day 1, n=15
  Interventions: Biological: BPZE1
- Group 3 (Placebo Comparator): 800 microliters of Placebo administered intranasally with the VaxINator device on Day 1, n=15
  Interventions: Other: Placebo
- Group 4 (Experimental): 800 microliters (10^9 CFU) of BPZE1 administered intranasally with a needleless tuberculin syringe on Day 1, n=5
  Interventions: Biological: BPZE1

INTERVENTIONS:
Biological: BPZE1 — Lyophilized, live-attenuated Bordetella pertussis vaccine reconstituted with sterile water for injection (SWFI) and administered as a single intranasal dose of either 10^7 colony forming units (CFU) or 10^9 CFU.
  Arms: Group 1; Group 2; Group 4
Other: Placebo — The placebo consists of the same constituents in the same quantities as the BPZE1 investigational vaccines, absent the attenuated B. pertussis cells, reconstituted with sterile water for injection (SWFI).
  Arms: Group 3

SUMMARY:
This is a randomized, partially blind, placebo controlled, clinical trial evaluating a single intranasal dose of BPZE1 in healthy adults. The study will evaluate a lyophilized formulation of the product, with the goal of testing for the optimal dose for subsequent clinical trials. Fifty healthy adults, 18-49 years of age will be randomized to one of the four following treatment groups in a 3:3:3:1 ratio: 10^7 colony forming units (CFU) of BPZE1 administered by VaxINator device, 10^9 CFU of BPZE1 administered by VaxINator device, placebo administered by VaxINator device, 10^9 CFU of BPZE1 administered by needleless tuberculin syringe. Study duration will be approximately 12 months with a subject participation duration of approximately 6 months. The primary objective of this study is to assess the safety and tolerability of a single intranasal dose of either 10^7 or 10^9 CFU of lyophilized BPZE1 vaccine.

DETAILED DESCRIPTION:
This is a phase 2a, single center, randomized, partially blind, placebo controlled, clinical trial evaluating a single intranasal dose of either 10^7 colony forming units (CFU) or 10^9 CFU of BPZE1 in healthy adults. The study will evaluate a lyophilized formulation of the product, with the goal of testing for the optimal dose for subsequent clinical trials. Fifty healthy adults, 18-49 years of age will be randomized to one of the four following treatment groups in a 3:3:3:1 ratio: 10^7 CFU of BPZE1 administered by VaxINator device, 10^9 CFU of BPZE1 administered by VaxINator device, placebo administered by VaxINator device, 10^9 CFU of BPZE1 administered by needleless tuberculin syringe. Study duration will be approximately 12 months with a subject participation duration of approximately 6 months. The primary objective of this study is to assess the safety and tolerability of a single intranasal dose of either 10^7 or 10^9 CFU of lyophilized BPZE1 vaccine. The secondary objectives of this study are: 1) to assess the humoral immunogenicity of lyophilized BPZE1 vaccine at Day 15, Day 29 and Day 181 following receipt of one intranasal dose of 10^7 or 10^9 CFU of BPZE1; 2) to assess mucosal immunogenicity of lyophilized BPZE1 vaccine at Day 29 and Day 181 following receipt of one intranasal dose of 10^7 or 10^9 CFU of BPZE1; 3) to evaluate nasal clearance of BPZE1 by culture at Day 29 (and if still positive, at Day 46) following receipt of one intranasal dose of lyophilized BPZE1 vaccine of 10^7 or 10^9 CFU of BPZE1.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible to participate in this study must meet all inclusion criteria:

1. Provide written informed consent prior to initiation of any study procedures.
2. Able to understand and comply with planned study procedures and be available for all study visits.
3. Males or non-pregnant females, 18-49 years of age, inclusive.
4. In good health*.

   *As determined by medical history and physical examination to evaluate acute or currently ongoing chronic medical diagnoses or conditions, defined as those that have been present for at least 90 days that would affect the assessment of the safety of subjects or the immunogenicity of study vaccinations. Chronic medical diagnoses or conditions should be stable for the last 60 days. This includes no change in chronic prescription medication, dose, or frequency because of deterioration of the chronic medical diagnosis or condition in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, if it is in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition. Similarly, medication changes after enrollment and study vaccination are acceptable provided there was no deterioration in the subject's chronic medical condition that necessitated a medication change, and there is no additional risk to the subject or interference with the evaluation of responses to study vaccination. Note: Topical and inhaled medications (with the exception of inhaled or nasal corticosteroids within 30 days prior to enrollment), herbals, vitamins, and supplements are permitted.
5. Oral temperature is < / = 100 degrees Fahrenheit.
6. Pulse is 45 to 100 bpm, inclusive*. *Pulse can be 45 to 50 bpm, inclusive, if no other symptoms are present. Otherwise, pulse should be 50-100 bpm.
7. Systolic blood pressure is 85 to 150 mm Hg, inclusive.
8. Diastolic blood pressure is 55 to 95 mm Hg, inclusive.
9. White blood cell count is 3,900 cells/microliter or greater*.

   *Abnormalities in white blood count, hemoglobin, platelet count, alanine aminotransferase, and serum creatinine that are suspected to be due to laboratory anomalies may be repeated once to ensure accuracy; additionally, otherwise eligible subjects with grade 1 abnormalities in these values may be considered for enrollment if, in the opinion of the investigator (or clinician on the 1572), the abnormalities are not clinically significant and do not pose additional risk to the study or the volunteer.
10. Hemoglobin is 13.0 g/dL or greater (men) or 11.8 g/dL or greater (women)*. *Abnormalities in white blood count, hemoglobin, platelet count, alanine aminotransferase, and serum creatinine that are suspected to be due to laboratory anomalies may be repeated once to ensure accuracy; additionally, otherwise eligible subjects with grade 1 abnormalities in these values may be considered for enrollment if, in the opinion of the investigator (or clinician on the 1572), the abnormalities are not clinically significant and do not pose additional risk to the study or the volunteer.
11. Platelet count is 135,000 cells/microliter or greater*.

    *Abnormalities in white blood count, hemoglobin, platelet count, alanine aminotransferase, and serum creatinine that are suspected to be due to laboratory anomalies may be repeated once to ensure accuracy; additionally, otherwise eligible subjects with grade 1 abnormalities in these values may be considered for enrollment if, in the opinion of the investigator (or clinician on the 1572), the abnormalities are not clinically significant and do not pose additional risk to the study or the volunteer.
12. Alanine aminotransferase is < 45 U/L (women) or 62 U/L (men)*.

    *Abnormalities in white blood count, hemoglobin, platelet count, alanine aminotransferase, and serum creatinine that are suspected to be due to laboratory anomalies may be repeated once to ensure accuracy; additionally, otherwise eligible subjects with grade 1 abnormalities in these values may be considered for enrollment if, in the opinion of the investigator (or clinician on the 1572), the abnormalities are not clinically significant and do not pose additional risk to the study or the volunteer.
13. Serum creatinine is < / = 1.25 mg/dL (men) or 1.11 mg/dL (women)*.

    *Abnormalities in white blood count, hemoglobin, platelet count, alanine aminotransferase, and serum creatinine that are suspected to be due to laboratory anomalies may be repeated once to ensure accuracy; additionally, otherwise eligible subjects with grade 1 abnormalities in these values may be considered for enrollment if, in the opinion of the investigator (or clinician on the 1572), the abnormalities are not clinically significant and do not pose additional risk to the study or the volunteer.
14. Negative serum HIV antibody assay.
15. Women of childbearing potential* must use an acceptable contraception method** from 30 days before study vaccination until 60 days after vaccination.

    *Not sterilized via tubal ligation, bilateral oophorectomy, salpingectomy, hysterectomy, or successful Essure(R) placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or < 1 year has passed since the last menses if menopausal.
    * Includes non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more prior to the subject receiving study vaccination, barrier methods such as condoms or diaphragms/cervical caps with spermicide, effective intrauterine devices, NuvaRing(R), and licensed hormonal methods such as implants, injectables or oral contraceptives ("the pill").
16. Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to study vaccination.

Exclusion Criteria:

1. Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
2. Have known or suspected active chronic autoinflammatory condition.
3. Have known active neoplastic disease (excluding non-melanoma skin cancer) or a history of any hematologic malignancy.
4. Have a history of persistent asthma, major anatomic nasopharyngeal abnormality, or sinus polyp disease due to chronic sinusitis*.

   *If a patient has a history of nasopharyngeal surgery such as, but not limited to rhinoplasty, tonsillectomy or sinus surgery, adequate healing time per the judgement of the investigator must occur prior to enrollment.
5. Have known hepatitis B or hepatitis C infection.
6. Have a history of alcohol or drug abuse within 5 years prior to study vaccination.
7. Currently untreated or clinically unstable (in the opinion of the investigator) schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
8. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 5 years prior to study vaccination.
9. Have received corticosteroids (including oral, parenteral, inhaled, nasal, or intra-articular) of any dose within 30 days prior to study vaccination.
10. Individual with PT serum IgG antibodies > / = 20 IU/mL and / or PRN serum IgG antibodies > / = 125 IU/ml.
11. Unwilling to refrain from smoking tobacco for 28 days post vaccination.
12. Receipt of immunoglobulin or blood derived products within 90 days of enrollment.
13. Receipt of a vaccine against pertussis in the past 2 years.
14. Receipt of a live vaccine within 30 days of study vaccination or an inactivated vaccine within 14 days of study vaccination.
15. Planned vaccination with a licensed vaccine within 28 days of study vaccination.
16. History of severe allergic reaction (e.g., anaphylaxis) or Bell's palsy, or Guillain-Barre syndrome, after a previous dose of any diphtheria toxoid-tetanus toxoid-, or pertussis-containing vaccine, or encephalopathy within 7 days of administration of a previous pertussis containing vaccine.
17. History of a progressive neurologic disorder.
18. In close contact* with children less than 1 year of age or contact with persons with known immunocompromising conditions.

    *Close contact includes sharing a household, serving as a healthcare worker, or working professionally in settings with repeated exposures.
19. Receipt of B. pertussis-active antibiotics* within 7 days prior to vaccination.

    *B. pertussis active antibiotics include macrolides, fluoroquinolones, trimethoprim-sulfamethoxazole, tetracyclines.
20. Known hypersensitivity to any component of the study vaccine.
21. Hypersensitivity to azithromycin, which may be used in the event of ongoing BPZE1 colonization.
22. Any condition that, in the opinion of the investigator, might interfere with objectives of the study or safety to the individual.
23. Acute illness, including temperature > 100 degrees Fahrenheit within one week prior to vaccination*.

    * Enrollment may be postponed if acute illness occurs; subjects must remain within the screening window, however, and must be rescreened if > 30 days elapses prior to enrollment.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population includes 50 healthy adults,18-49 years of age, inclusive, who meet all eligibility criteria. Participants were enrolled between 01NOV2018 and 06DEC2019.
Groups:
- BPZE1 10^7 CFU by VaxINator: 800 microliters (10^7 CFU) of B. pertussis vaccine (BPZE1) administered intranasally with the VaxINator device on Day 1.
  BPZE1: Lyophilized, live-attenuated Bordetella pertussis vaccine reconstituted with sterile water for injection (SWFI) and administered as a single intranasal dose of 10^7 colony forming units (CFU).
- BPZE1 10^9 CFU by VaxINator: 800 microliters (10^9 CFU) of BPZE1 administered intranasally with the VaxINator device on Day 1.
  BPZE1: Lyophilized, live-attenuated Bordetella pertussis vaccine reconstituted with sterile water for injection (SWFI) and administered as a single intranasal dose of 10^9 colony forming units (CFU).
- BPZE1 10^9 CFU by Syringe: 800 microliters (10^9 CFU) of BPZE1 administered intranasally with a needleless tuberculin syringe on Day 1.
  BPZE1: Lyophilized, live-attenuated Bordetella pertussis vaccine reconstituted with sterile water for injection (SWFI) and administered as a single intranasal dose of 10^9 colony forming units (CFU) .
- Placebo by VaxINator: 800 microliters of Placebo administered intranasally with the VaxINator device on Day 1.
  Placebo: The placebo consists of the same constituents in the same quantities as the BPZE1 investigational vaccines, absent the attenuated B. pertussis cells, reconstituted with sterile water for injection (SWFI).
Period: Overall Study
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Started | 15 | 15 | 5 | 15
Completed | 15 | 15 | 5 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study population includes 50 healthy adults, 18-49 years of age, inclusive, who meet all eligibility criteria.
Groups:
- BPZE1 10^7 CFU by VaxINator: 800 microliters (10^7 CFU) of BPZE1 administered intranasally with the VaxINator device on Day 1.
- BPZE1 10^9 CFU by VaxINator: 800 microliters (10^9 CFU) of BPZE1 administered intranasally with the VaxINator device on Day 1.
- BPZE1 10^9 CFU by Syringe: 800 microliters (10^9 CFU) of BPZE1 administered intranasally with a needleless tuberculin syringe on Day 1.
- Placebo by VaxINator: 800 microliters of Placebo administered intranasally with the VaxINator device on Day 1.
- Total: Total of all reporting groups
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator | Total
Number analyzed (Participants) | 15 | 15 | 5 | 15 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (10.7) | 29.1 (8.8) | 30.2 (8.9) | 30.9 (9.5) | 30.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 2 | 11 | 31
  Male | 6 | 6 | 3 | 4 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 15 | 15 | 5 | 14 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 1 | 0 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 10 | 14 | 5 | 13 | 42
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events of Special Interest (AESIs)
Description: AESIs included medically attended wheezing events given the route of study product administration and the nature of the study product.
Time Frame: Day 1 through Day 29
Population: The safety population consists of all participants who received the study vaccine and for whom any data on safety were available.
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Experiencing New Onset Chronic Medical Conditions (NOCMCs)
Description: NOCMCs are defined as new medical conditions, not present at the time of screening or enrollment, that require ongoing medical care and intervention.
Time Frame: Day 1 through Day 181
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
Participants | 1 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Experiencing Serious Adverse Events (SAEs)
Description: An adverse event was considered serious if, in the view of either the site principal investigator or sponsor, it resulted in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect, or, when, based upon appropriate medical judgment they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Day 1 through Day 181
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Experiencing Solicited Local Reactogenicity Adverse Events (AEs)
Description: The solicited local reactogenicity events included runny nose, stuffy nose/congestion, nasal pain/irritation, epistaxis, sneezing, sinus pressure/pain, sore/irritated throat, cough, and shortness of breath/wheezing.
Time Frame: Day 1 through Day 15
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
Participants
  Runny nose | 6 | 7 | 2 | 5
  Stuffy nose/congestion | 8 | 8 | 2 | 6
  Nasal pain/irritation | 1 | 1 | 0 | 0
  Epistaxis | 1 | 0 | 0 | 1
  Sneezing | 4 | 5 | 1 | 3
  Sinus pressure/pain | 1 | 4 | 0 | 2
  Sore/irritated throat | 4 | 4 | 2 | 3
  Cough | 6 | 2 | 2 | 2
  Shortness of breath/wheezing | 2 | 1 | 0 | 0

5. Primary Outcome: Number of Participants Experiencing Solicited Systemic Reactogenicity AEs
Description: The solicited systemic reactogenicity events included fever, feverishness, fatigue, malaise, myalgia, arthralgia, headache, and rash/hypersensitivity.
Time Frame: Day 1 through Day 15
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
Participants
  Fever | 1 | 0 | 0 | 0
  Feverishness | 1 | 2 | 0 | 1
  Fatigue (tiredness) | 4 | 4 | 2 | 5
  Malaise (general unwell feeling) | 3 | 3 | 1 | 2
  Myalgia (body aches/muscular pain) | 0 | 2 | 1 | 1
  Arthralgia (joint pain) | 0 | 3 | 1 | 1
  Headache | 5 | 9 | 2 | 8
  Rash/hypersensitivity | 1 | 0 | 0 | 0

6. Primary Outcome: Number of Participants Experiencing Unsolicited Non-Serious AEs
Description: Adverse events were defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. Unsolicited non-serious AEs were documented and reported from the time of vaccination through Day 29.
Time Frame: Day 1 through Day 29
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
Participants | 3 | 3 | 1 | 5

7. Primary Outcome: Number of Participants Experiencing Severe Solicited Local Reactogenicity Adverse Events
Description: Solicited local reactogenicity events include runny nose, stuffy nose/congestion, nasal pain/irritation, epistaxis, sneezing, sinus pressure/pain, sore/irritated throat, cough, and shortness of breath/wheezing. They were graded as grade 1 (mild), grade 2 (moderate), or grade 3 (severe). Severe local events were those that required medical care or caused significant discomfort that prevented daily activity, including sore/irritated throat preventing eating or drinking and cough preventing sleep. Severe epistaxis events were bleeding events that required a medical encounter. Severe stuffy nose/congestion events caused the participant to be unable to breathe through the nose or to seek medical care.
Time Frame: Day 1 through Day 15
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
Participants
  Runny nose | 0 | 0 | 0 | 0
  Stuffy nose/congestion | 0 | 0 | 0 | 0
  Nasal pain/irritation | 0 | 0 | 0 | 0
  Epistaxis | 0 | 0 | 0 | 0
  Sneezing | 0 | 0 | 0 | 0
  Sinus pressure/pain | 0 | 0 | 0 | 0
  Sore/irritated throat | 0 | 0 | 0 | 0
  Cough | 0 | 0 | 0 | 0
  Shortness of breath/wheezing | 0 | 0 | 0 | 0

8. Secondary Outcome: Geometric Mean Fold Rise From Screening of the Ratio of Filamentous Hemagglutinin-specific IgA (FHA-IgA) to Total IgA by Nasal Aspirate
Description: Nasal aspirate samples were collected from all participants at screening (baseline), Day 29, and Day 181 to measure total mucosal IgA levels via ELISA assay and mucosal IgA levels to filamentous hemagglutinin (FHA) pertussis antigen via a bead-based assay. Total mucosal IgA levels were reported in µg/mL; antigen-specific IgA results were reported in ELISA units/mL.
  The ratio of FHA-IgA to total mucosal IgA was computed for each participant at each time point, and the fold rise from baseline of this ratio was subsequently calculated for each participant. The geometric mean fold rise of the ratio was calculated for each study arm.
Time Frame: Screening, Day 29, Day 181
Population: The Immunogenicity Population includes all participants who received the study vaccination and contributed both pre-vaccination samples and either at least one post vaccination sample for humoral immunogenicity testing for which results were reported, or at least one post vaccination nasal sample for which results were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
fold rise
  Day 29 | 1.2 [0.8 to 1.7] | 1.7 [1.0 to 3.0] | 0.3 [0 to 10.3] | 1 [0.7 to 1.6]
  Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  Day 181 | 0.8 [0.5 to 1.3] | 2 [1.2 to 3.3] | 0.4 [0 to 10.1] | 1.2 [0.7 to 2.1]

9. Secondary Outcome: Geometric Mean Fold Rise From Screening of the Ratio of Fimbriae-Specific IgA (FIM-IgA) to Total IgA by Nasal Aspirate
Description: Nasal aspirate samples were collected from all participants at screening (baseline), Day 29, and Day 181 to measure total mucosal IgA levels via ELISA assay and mucosal IgA levels to fimbriae 2/3 (FIM) pertussis antigen via a bead-based assay. Total mucosal IgA levels were reported in µg/mL; antigen-specific IgA results were reported in ELISA units/mL.
  The ratio of FIM-IgA to total mucosal IgA was computed for each participant at each time point, and the fold rise from baseline of this ratio was subsequently calculated for each participant. The geometric mean fold rise of the ratio was calculated for each study arm.
Time Frame: Screening, Day 29, and Day 181
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
fold rise
  Day 29 | 1.7 [0.7 to 3.8] | 6.2 [2.2 to 17.3] | 0.7 [0 to 36.3] | 0.6 [0.3 to 1.4]
  Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  Day 181 | 1.1 [0.6 to 1.9] | 6.7 [2.8 to 16.0] | 1 [0.1 to 18.9] | 0.8 [0.3 to 1.9]

10. Secondary Outcome: Geometric Mean Fold Rise From Screening of the Ratio of Pertactin-Specific IgA (PRN-IgA) to Total IgA by Nasal Aspirate
Description: Nasal aspirate samples were collected from all participants at screening (baseline), Day 29, and Day 181 to measure total mucosal IgA levels via ELISA assay and mucosal IgA levels to pertactin (PRN) pertussis antigen via a bead-based assay. Total mucosal IgA levels were reported in µg/mL; antigen-specific IgA results were reported in ELISA units/mL.
  The ratio of PRN-IgA to total mucosal IgA was computed for each participant at each time point, and the fold rise from baseline of this ratio was subsequently calculated for each participant. The geometric mean fold rise of the ratio was calculated for each study arm.
Time Frame: Screening, Day 29, and Day 181
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
fold rise
  Day 29 | 1.1 [0.8 to 1.5] | 3.3 [1.3 to 8.3] | 1.3 [0.1 to 27.0] | 0.8 [0.5 to 1.3]
  Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  Day 181 | 1.1 [0.8 to 1.5] | 3.5 [1.4 to 8.8] | 3.3 [1.0 to 10.5] | 1 [0.5 to 1.9]

11. Secondary Outcome: Geometric Mean Fold Rise From Screening of the Ratio of Pertussis Toxin-Specific IgA (PT-IgA) to Total IgA by Nasal Aspirate
Description: Nasal aspirate samples were collected from all participants at screening (baseline), Day 29, and Day 181 to measure total mucosal IgA levels via ELISA assay and mucosal IgA levels to pertussis toxin (PT) pertussis antigen via a bead-based assay. Total mucosal IgA levels were reported in µg/mL; antigen-specific IgA results were reported in ELISA units/mL.
  The ratio of PT-IgA to total mucosal IgA was computed for each participant at each time point, and the fold rise from baseline of this ratio was subsequently calculated for each participant. The geometric mean fold rise of the ratio was calculated for each study arm.
Time Frame: Screening, Day 29, and Day 181
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
fold rise
  Day 29 | 0.9 [0.5 to 1.5] | 1.4 [0.8 to 2.5] | 0.9 [0.4 to 2.0] | 2.2 [1.4 to 3.5]
  Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  Day 181 | 1.3 [0.8 to 1.9] | 1.6 [0.9 to 2.6] | 1.6 [0.7 to 3.7] | 1.2 [0.7 to 2.2]

12. Secondary Outcome: Geometric Mean Fold Rise From Baseline Serum IgA and Serum IgG ELISA Titers to Filamentous Hemagglutinin (FHA)
Description: Approximately 10 mL of venous blood was collected from participants immediately prior to the first study vaccination on Day 1 (baseline), Day 15, Day 29, and Day 181 to perform a bead-based assay to measure serum IgA and serum IgG levels (in ELISA units/mL) to filamentous hemagglutinin (FHA) pertussis antigen.
  The fold rise in FHA-IgA from baseline was calculated for each participant and the geometric mean of the fold rise was calculated for each study arm.
Time Frame: Day 1, Day 15, Day 29, and Day 181
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
fold rise
  IgA - Day 15 | 0.8 [0.4 to 1.4] | 1.3 [0.9 to 2.0] | 1.4 [0.7 to 2.8] | 1 [0.6 to 1.5]
  IgA - Day 29 | 1.4 [0.5 to 3.5] | 2.5 [1.3 to 4.6] | 3 [0.5 to 17.6] | 0.8 [0.6 to 1.1]
  IgA - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgA - Day 181 | 1.2 [0.5 to 3.2] | 2.1 [1.2 to 3.6] | 2.3 [0.5 to 10] | 1.1 [0.6 to 2.0]
  IgG - Day 15 | 1 [0.8 to 1.3] | 1.2 [0.8 to 1.7] | 0.8 [0.4 to 1.4] | 1.1 [0.9 to 1.4]
  IgG - Day 29 | 1.7 [0.8 to 3.8] | 1.5 [1.0 to 2.3] | 1.3 [0.4 to 4.2] | 0.9 [0.8 to 1.1]
  IgG - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgG - Day 181 | 1.8 [0.9 to 3.8] | 1.7 [1.1 to 2.5] | 1.2 [0.7 to 2.1] | 1 [0.7 to 1.4]

13. Secondary Outcome: Geometric Mean Fold Rise From Baseline of Serum IgA and Serum IgG ELISA Titers to Fimbriae 2/3 (FIM)
Description: Approximately 10 mL of venous blood was collected from participants immediately prior to the first study vaccination on Day 1 (baseline), Day 15, Day 29, and Day 181 to perform a bead-based assay to measure serum IgA levels and serum IgG levels (in ELISA units/mL) to fimbriae 2/3 (FIM) pertussis antigen.
  The fold rise in FIM-IgA and FIM-IgG from baseline was calculated for each participant and the geometric mean of the fold rise was calculated for each study arm.
Time Frame: Day 1, Day 15, Day 29, and Day 181
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
fold rise
  IgA - Day 15 | 1 [0.8 to 1.2] | 1.1 [0.6 to 1.8] | 1.1 [0.9 to 1.4] | 1 [0.8 to 1.2]
  IgA - Day 29 | 2.1 [0.8 to 5.4] | 2.2 [0.9 to 5.3] | 3.2 [0.4 to 26.8] | 0.7 [0.4 to 1.3]
  IgA - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgA - Day 181 | 1.4 [0.7 to 2.7] | 2 [0.9 to 4.7] | 2.3 [0.4 to 13.4] | 1.1 [0.8 to 1.5]
  IgG - Day 15 | 1.1 [0.9 to 1.3] | 1.5 [1.0 to 2.3] | 1 [0.6 to 1.6] | 1 [0.8 to 1.4]
  IgG - Day 29 | 1.6 [0.8 to 3.2] | 2.6 [1.3 to 5.3] | 1.2 [0.8 to 2.0] | 1 [0.9 to 1.2]
  IgG - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgG - Day 181 | 1.2 [0.9 to 1.6] | 2.8 [1.3 to 6.0] | 1.2 [1.0 to 1.6] | 0.9 [0.7 to 1.2]

14. Secondary Outcome: Geometric Mean Fold Rise From Baseline of Serum IgA and Serum IgG ELISA Titers to Pertactin (PRN)
Description: Approximately 10 mL of venous blood was collected from participants immediately prior to the first study vaccination on Day 1 (baseline), Day 15, Day 29, and Day 181 to perform a bead-based assay to measure serum IgA and serum IgG levels (in ELISA units/mL) to pertactin (PRN) pertussis antigen.
  The fold rise in PRN-IgA and PRN-IgG from baseline was calculated for each participant and the geometric mean of the fold rise was calculated for each study arm.
Time Frame: Day 1, Day 15, Day 29, and Day 181
Population: The Immunogenicity Population includes all participants who have received the study vaccination and contributed both pre-vaccination samples and either at least one post vaccination sample for humoral immunogenicity testing for which results were reported, or at least one post vaccination nasal sample for which results were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
fold rise
  IgA - Day 15 | 0.7 [0.5 to 1.0] | 1.6 [1.2 to 2.3] | 1.1 [0.6 to 2.3] | 1.1 [0.8 to 1.5]
  IgA - Day 29 | 0.9 [0.4 to 1.8] | 3.2 [1.9 to 5.7] | 2.2 [0.6 to 8.1] | 1.1 [0.8 to 1.6]
  IgA - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgA - Day 181 | 0.9 [0.4 to 1.7] | 3.2 [2.1 to 4.9] | 1.5 [0.4 to 5.4] | 1.3 [0.9 to 1.8]
  IgG - Day 15 | 1 [0.7 to 1.4] | 1.5 [1.1 to 2.1] | 0.9 [0.5 to 1.4] | 1.1 [0.8 to 1.6]
  IgG - Day 29 | 1.7 [0.7 to 4.0] | 2.3 [1.3 to 4.3] | 1.2 [0.4 to 3.2] | 0.9 [0.7 to 1.1]
  IgG - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgG - Day 181 | 1.5 [0.5 to 4.2] | 2.5 [1.5 to 4.3] | 0.9 [0.3 to 2.3] | 0.9 [0.7 to 1.2]

15. Secondary Outcome: Geometric Mean Fold Rise From Baseline of Serum IgA and Serum IgG ELISA Titers to Pertussis Toxin (PT)
Description: Approximately 10 mL of venous blood was collected from participants immediately prior to the first study vaccination on Day 1 (baseline), Day 15, Day 29, and Day 181 to perform a bead-based assay to measure serum IgA and serum IgG levels (in ELISA units/mL) to pertussis toxin (PT) pertussis antigen.
  The fold rise in PT-IgA and PT-IgG from baseline was calculated for each participant and the geometric mean of the fold rise was calculated for each study arm.
Time Frame: Day 1, Day 15, Day 29, and Day 181
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
fold rise
  IgA - Day 15 | 1.3 [0.8 to 2.1] | 1.9 [0.8 to 4.3] | 1 [0.5 to 1.9] | 1 [0.4 to 2.1]
  IgA - Day 29 | 1.4 [0.7 to 2.8] | 1.9 [1.1 to 3.6] | 1.4 [0.3 to 6.6] | 1.2 [0.5 to 2.7]
  IgA - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgA - Day 181 | 1 [0.5 to 2.2] | 1.8 [1.2 to 2.7] | 1 [0.3 to 3.2] | 1.4 [0.8 to 2.6]
  IgG - Day 15 | 1.1 [0.8 to 1.4] | 1.2 [0.9 to 1.6] | 0.7 [0.4 to 1.3] | 1 [0.8 to 1.3]
  IgG - Day 29 | 1.5 [0.6 to 3.9] | 1.4 [0.9 to 1.9] | 1.5 [0.3 to 7.8] | 1 [0.8 to 1.2]
  IgG - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgG - Day 181 | 1.9 [0.7 to 5.3] | 1.4 [1.0 to 2.0] | 1.1 [0.4 to 3.0] | 0.9 [0.7 to 1.1]

16. Secondary Outcome: Geometric Mean Titer by Serum IgA and Serum IgG to Fimbriae 2/3
Description: Approximately 10 mL of venous blood was collected from participants immediately prior to the first study vaccination on Day 1 (baseline), Day 15, Day 29, and Day 181 to measure serum IgA and serum IgG levels (in ELISA units/mL) to fimbriae 2/3 (FIM) pertussis antigen via a bead-based assay. The geometric mean FIM-IgA titer and FIM-IgG titer were calculated for each study arm.
Time Frame: Day 1, Day 15, Day 29, and Day 181
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
titer
  IgA - Day 1 | 3.40 [1.64 to 7.04] | 3.94 [1.99 to 7.82] | 1.85 [0.34 to 10.17] | 2.68 [1.12 to 6.44]
  IgA - Day 15 | 3.27 [1.44 to 7.43] | 4.26 [2.05 to 8.89] | 2.04 [0.33 to 12.75] | 2.68 [1.06 to 6.77]
  IgA - Day 29 | 7.07 [2.30 to 21.73] | 8.84 [4.57 to 17.11] | 5.92 [1.17 to 29.86] | 1.79 [0.70 to 4.54]
  IgA - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgA - Day 181 | 5.30 [1.69 to 16.56] | 8.01 [4.35 to 14.76] | 4.29 [1.17 to 15.80] | 2.69 [1.08 to 6.70]
  IgG - Day 1 | 51.71 [21.47 to 124.54] | 15.98 [4.70 to 54.34] | 129.14 [33.05 to 504.51] | 24.48 [9.72 to 61.62]
  IgG - Day 15 | 56.73 [24.08 to 133.65] | 24.17 [8.59 to 68.04] | 129.80 [22.13 to 761.39] | 25.30 [9.27 to 69.07]
  IgG - Day 29 | 84.12 [33.20 to 213.14] | 41.30 [17.13 to 99.58] | 160.50 [39.43 to 653.35] | 24.35 [9.90 to 59.91]
  IgG - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgG - Day 181 | 80.27 [28.79 to 223.77] | 45.32 [20.61 to 99.69] | 159.90 [50.19 to 509.41] | 21.84 [7.45 to 64.00]

17. Secondary Outcome: Geometric Mean Titer by Serum IgA and Serum IgG to Pertactin
Description: Approximately 10 mL of venous blood was collected from participants immediately prior to the first study vaccination on Day 1 (baseline), Day 15, Day 29, and Day 181 to measure serum IgA levels and serum IgG levels (in ELISA units/mL) to pertactin (PRN) pertussis antigen via a bead-based assay. The geometric mean PRN-IgA titer and PRN-IgG titer were calculated for each study arm.
Time Frame: Day 1, Day 15, Day 29, and Day 181
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
titer
  IgA - Day 1 | 10.53 [5.78 to 19.18] | 3.82 [2.07 to 7.05] | 3.57 [0.36 to 35.49] | 2.88 [1.51 to 5.50]
  IgA - Day 15 | 7.69 [3.62 to 16.33] | 6.21 [3.67 to 10.51] | 4.07 [0.29 to 56.22] | 3.22 [1.54 to 6.74]
  IgA - Day 29 | 9.32 [3.80 to 22.87] | 12.38 [5.46 to 28.09] | 8.02 [0.80 to 80.35] | 3.19 [1.54 to 6.63]
  IgA - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgA - Day 181 | 7.90 [3.37 to 18.50] | 12.19 [5.88 to 25.26] | 5.43 [0.82 to 35.95] | 4.10 [1.90 to 8.85]
  IgG - Day 1 | 38.69 [17.89 to 83.67] | 17.68 [10.44 to 29.94] | 48.47 [10.30 to 228.02] | 8.81 [2.44 to 31.77]
  IgG - Day 15 | 38.59 [20.87 to 71.36] | 26.42 [16.67 to 41.88] | 41.42 [13.35 to 128.47] | 9.58 [3.00 to 30.62]
  IgG - Day 29 | 65.11 [35.36 to 119.90] | 41.07 [23.18 to 72.76] | 58.20 [23.31 to 145.33] | 7.63 [2.13 to 27.30]
  IgG - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgG - Day 181 | 53.49 [24.22 to 118.15] | 44.92 [28.07 to 71.89] | 42.76 [9.37 to 195.09] | 11.36 [3.70 to 34.88]

18. Secondary Outcome: Geometric Mean Titer by Serum IgA and Serum IgG to Pertussis Toxin
Description: Approximately 10 mL of venous blood was collected from participants immediately prior to the first study vaccination on Day 1 (baseline), Day 15, Day 29, and Day 181 to measure serum IgA levels and serum IgG levels (in ELISA units/mL) to pertussis toxin (PT) pertussis antigen via a bead-based assay. The geometric mean PT-IgA titer and PT-IgG titer were calculated for each study arm.
Time Frame: Day 1, Day 15, Day 29, and Day 181
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
titer
  IgA - Day 1 | 0.66 [0.38 to 1.15] | 0.48 [0.24 to 0.98] | 0.91 [0.15 to 5.53] | 0.82 [0.36 to 1.88]
  IgA - Day 15 | 0.86 [0.45 to 1.65] | 0.92 [0.44 to 1.93] | 0.88 [0.24 to 3.16] | 0.80 [0.51 to 1.25]
  IgA - Day 29 | 0.91 [0.47 to 1.77] | 0.95 [0.52 to 1.71] | 1.29 [0.30 to 5.47] | 0.99 [0.54 to 1.81]
  IgA - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgA - Day 181 | 0.82 [0.41 to 1.62] | 0.86 [0.57 to 1.28] | 0.91 [0.21 to 3.92] | 1.28 [0.75 to 2.18]
  IgG - Day 1 | 3.36 [1.73 to 6.53] | 4.00 [1.73 to 9.27] | 10.10 [1.33 to 76.89] | 3.41 [1.51 to 7.71]
  IgG - Day 15 | 3.65 [1.82 to 7.30] | 4.77 [2.43 to 9.37] | 7.36 [1.47 to 36.78] | 3.38 [1.37 to 8.34]
  IgG - Day 29 | 5.20 [2.25 to 12.05] | 5.41 [2.49 to 11.79] | 15.01 [2.52 to 89.24] | 3.42 [1.45 to 8.07]
  IgG - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgG - Day 181 | 6.39 [2.60 to 15.70] | 5.67 [2.81 to 11.47] | 10.86 [1.67 to 70.71] | 3.09 [1.19 to 8.03]

19. Secondary Outcome: Percentage of Participants Achieving Seroconversion to One or More Pertussis Antigens as Measured by Serum IgA or Serum IgG Levels
Description: Approximately 10 mL of venous blood was collected from participants immediately prior to the first study vaccination on Day 1 (baseline), Day 15, Day 29, and Day 181 to measure via a bead-based assay serum IgA and serum IgG levels (in ELISA units/mL) to pertussis toxin, filamentous hemagglutinin, pertactin, and fimbriae 2/3 pertussis antigens.
  Seroconversion was defined as at least a 2-fold rise in antigen-specific IgA or antigen-specific IgG levels post-baseline compared to baseline levels. The percentage of participants who seroconverted to at least one pertussis antigen at each and across immunogenicity timepoints (Day 15, Day 29, and Day 181) was calculated.
Time Frame: Day 15, Day 29, and Day 181
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
percentage of participants
  Any Time Point | 67 [38.4 to 88.2] | 100 [78.2 to 100] | 60 [14.7 to 94.7] | 73 [44.9 to 92.2]
  Day 15 | 33 [11.8 to 61.6] | 67 [38.4 to 88.2] | 60 [14.7 to 94.7] | 40 [16.3 to 67.7]
  Day 29 | 53 [26.6 to 78.7] | 93 [68.1 to 99.8] | 60 [14.7 to 94.7] | 47 [21.3 to 73.4]
  Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  Day 181 | 42 [15.2 to 72.3] | 93 [68.1 to 99.8] | 60 [14.7 to 94.7] | 57 [28.9 to 82.3]
Statistical Analysis 1: Comparison: BPZE1 10^7 CFU by VaxINator vs Placebo by VaxINator; At any time point; Test type: Superiority; p = 0.807, Barnard's exact test
Statistical Analysis 2: Comparison: BPZE1 10^9 CFU by VaxINator vs Placebo by VaxINator; At any time point; Test type: Superiority; p = 0.043, Barnard's exact test

20. Secondary Outcome: Percentage of Participants Achieving Seroconversion to Two or More Pertussis Antigens as Measured by Serum IgA or Serum IgG Levels
Description: Approximately 10 mL of venous blood was collected from participants immediately prior to the first study vaccination on Day 1 (baseline), Day 15, Day 29, and Day 181 to measure via a bead-based assay serum IgA and serum IgG levels (in ELISA units/mL) to pertussis toxin, filamentous hemagglutinin, pertactin, and fimbriae 2/3 pertussis antigens.
  Seroconversion was defined as at least a 2-fold rise in antigen-specific IgA levels or antigen-specific IgG levels post-baseline compared to baseline levels. The percentage of participants who seroconverted to at least two pertussis antigens at each and across all immunogenicity timepoints (Day 15, Day 29, and Day 181) was calculated.
Time Frame: Day 15, Day 29, and Day 181
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
percentage of participants
  Any Time Point | 53 [26.6 to 78.7] | 73 [44.9 to 92.2] | 60 [14.7 to 94.7] | 53 [26.6 to 78.7]
  Day 15 | 7 [0.2 to 31.9] | 53 [26.6 to 78.7] | 20 [0.5 to 71.6] | 27 [7.8 to 55.1]
  Day 29 | 27 [7.8 to 55.1] | 73 [44.9 to 92.2] | 60 [14.7 to 94.7] | 20 [4.3 to 48.1]
  Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  Day 181 | 25 [5.5 to 57.2] | 67 [38.4 to 88.2] | 60 [14.7 to 94.7] | 36 [12.8 to 64.9]
Statistical Analysis 1: Comparison: BPZE1 10^7 CFU by VaxINator vs Placebo by VaxINator; Any time point; Test type: Superiority; p = 1.000, Barnard's exact test
Statistical Analysis 2: Comparison: BPZE1 10^9 CFU by VaxINator vs Placebo by VaxINator; Any time point; Test type: Superiority; p = 0.301, Barnard's exact test

21. Secondary Outcome: Percentage of Participants Achieving Seroconversion to One or More Pertussis Antigens as Measured by the Ratio of Antigen-Specific Mucosal IgA Levels to Total Mucosal IgA Levels
Description: Nasal aspirate samples were collected from all participants at screening (baseline), Day 29, and Day 181 to measure total mucosal IgA levels via ELISA assay and mucosal IgA levels to pertussis vaccine antigens via a bead-based assay. Total mucosal IgA levels were reported in µg/mL; antigen-specific IgA results were reported in ELISA units/mL.
  The titer ratio of antigen-specific IgA to total mucosal IgA was computed for each participant at each time point, and the fold rise from baseline of this ratio was subsequently calculated for each participant.
  Seroconversion was defined as at least a 2-fold rise in antigen-specific titer ratios post-baseline compared to baseline titer ratios. The percentage of participants who seroconverted to at least one pertussis antigen at each and any immunogenicity timepoint was calculated.
Time Frame: Day 29 and Day 181
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
percentage of participants
  Any Time Point | 60 [32.3 to 83.7] | 93 [68.1 to 99.8] | 80 [28.4 to 99.5] | 80 [51.9 to 95.7]
  Day 29 | 53 [26.6 to 78.7] | 73 [44.9 to 92.2] | 60 [14.7 to 94.7] | 73 [44.9 to 92.2]
  Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  Day 181 | 50 [21.1 to 78.9] | 93 [68.1 to 99.8] | 80 [28.4 to 99.5] | 50 [23.0 to 77.0]
Statistical Analysis 1: Comparison: BPZE1 10^7 CFU by VaxINator; Any time point; Test type: Superiority; p = 1.000, Barnard's exact test
Statistical Analysis 2: Comparison: BPZE1 10^9 CFU by VaxINator vs Placebo by VaxINator; Any time point; Test type: Superiority; p = 0.009, Barnard's exact test

22. Secondary Outcome: Percentage of Participants With Detectable B. Pertussis From Nasopharyngeal Cultures
Description: Colonization of live B. pertussis organism was assessed from a nasopharyngeal swab performed 28 days after vaccine administration (Day 29) to ensure all participants were cleared of colonization. Standard microbiologic techniques were used to assess the presence of B. pertussis by culture.
  If any participants were positive for B. pertussis culture at Day 29, they were asked to return at Day 46 for a repeat culture. If the participant was not positive for B. pertussis at Day 29, no subsequent nasopharyngeal samples for culture were collected.
Time Frame: Day 29 and Day 46
Population: The Per Protocol (PP) Population includes all participants in the immunogenicity population, excluding participants ineligible at baseline. Data is excluded from PP analyses from visits after major protocol deviations and study visits that occurred greater than 3 days out of window. Data from 1 participant was excluded from the BPZE1 10^7 CFU by VaxINator group due to receipt of immunosuppressive therapy within 30 days of study vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 14 | 15 | 5 | 15
percentage of participants
  Day 29 | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 52.2] | 0 [0.0 to 21.8]
  Day 46: number analyzed (Participants) | 0 | 0 | 0 | 0

23. Secondary Outcome: Percentage of Participants Achieving Seroconversion to Filamentous Hemagglutinin as Measured by Serum IgA and Serum IgG Levels
Description: Approximately 10 mL of venous blood was collected from participants immediately prior to the first study vaccination on Day 1 (baseline), Day 15, Day 29, and Day 181 to measure via a bead-based assay serum IgA levels and serum IgG levels (in ELISA units/mL) to filamentous hemagglutinin (FHA) pertussis antigen.
  Seroconversion was defined as at least a 2-fold rise in antigen-specific IgA and IgG levels post-baseline compared to baseline levels. The percentage of participants who seroconverted to FHA-IgA and FHA-IgG at any and each immunogenicity timepoint (Day 15, Day 29, and Day 181) was calculated.
Time Frame: Day 15, Day 29, and Day 181
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
percentage of participants
  IgA - Any Time Point | 20 [4.3 to 48.1] | 67 [38.4 to 88.2] | 60 [14.7 to 94.7] | 33 [11.8 to 61.6]
  IgA - Day 15 | 13 [1.7 to 40.5] | 20 [4.3 to 48.1] | 40 [5.3 to 85.3] | 7 [0.2 to 31.9]
  IgA - Day 29 | 13 [1.7 to 40.5] | 67 [38.4 to 88.2] | 60 [14.7 to 94.7] | 7 [0.2 to 31.9]
  IgA - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgA - Day 181 | 17 [2.1 to 48.4] | 40 [16.3 to 67.7] | 60 [14.7 to 94.7] | 21 [4.7 to 50.8]
  IgG - Any Time Point | 47 [21.3 to 73.4] | 53 [26.6 to 78.7] | 40 [5.3 to 85.3] | 13 [1.7 to 40.5]
  IgG - Day 15 | 7 [0.2 to 31.9] | 7 [0.2 to 31.9] | 0 [0.0 to 52.2] | 7 [0.2 to 31.9]
  IgG - Day 29 | 33 [11.8 to 61.6] | 40 [16.3 to 67.7] | 40 [5.3 to 85.3] | 0 [0.0 to 21.8]
  IgG - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgG - Day 181 | 33 [9.9 to 65.1] | 47 [21.3 to 73.4] | 20 [0.5 to 71.6] | 7 [0.2 to 33.9]
Statistical Analysis 1: Comparison: BPZE1 10^7 CFU by VaxINator vs Placebo by VaxINator; IgA, any time point; Test type: Superiority; p = 0.526, Barnard's exact test
Statistical Analysis 2: Comparison: BPZE1 10^9 CFU by VaxINator vs Placebo by VaxINator; IgA, any time point; Test type: Superiority; p = 0.100, Barnard's exact test
Statistical Analysis 3: Comparison: BPZE1 10^7 CFU by VaxINator vs Placebo by VaxINator; IgG, any time point; Test type: Superiority; p = 0.055, Barnard's exact test
Statistical Analysis 4: Comparison: BPZE1 10^9 CFU by VaxINator vs Placebo by VaxINator; IgG, any time point; Test type: Superiority; p = 0.023, Barnard's exact test

24. Secondary Outcome: Percentage of Participants Achieving Seroconversion to Fimbriae 2/3 as Measured by Serum IgA and Serum IgG Levels
Description: Approximately 10 mL of venous blood was collected from participants immediately prior to the first study vaccination on Day 1 (baseline), Day 15, Day 29, and Day 181 to measure via a bead-based assay serum IgA and serum IgG levels (in ELISA units/mL) to fimbriae 2/3 (FIM) pertussis antigen.
  Seroconversion was defined as at least a 2-fold rise in antigen-specific IgA levels and IgG levels post-baseline compared to baseline levels. The percentage of participants who seroconverted to FIM-IgA or FIM-IgG at any and each immunogenicity timepoint (Day 15, Day 29, or and Day 181) was calculated.
Time Frame: Day 15, Day 29, and Day 181
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
percentage of participants
  IgA - Any Time Point | 27 [7.8 to 55.1] | 53 [26.6 to 78.7] | 60 [14.7 to 94.7] | 7 [0.2 to 31.9]
  IgA - Day 15 | 0 [0.0 to 21.8] | 13 [1.7 to 40.5] | 0 [0.0 to 52.2] | 0 [0.0 to 21.8]
  IgA - Day 29 | 27 [7.8 to 55.1] | 53 [26.6 to 78.7] | 60 [14.7 to 94.7] | 0 [0.0 to 21.8]
  IgA - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgA - Day 181 | 8 [0.2 to 38.5] | 40 [16.3 to 67.7] | 40 [5.3 to 85.3] | 7 [0.2 to 33.9]
  IgG - Any Time Point | 20 [4.3 to 48.1] | 53 [26.6 to 78.7] | 0 [0 to 52.2] | 13 [1.7 to 40.5]
  IgG - Day 15 | 0 [0.0 to 21.8] | 20 [4.3 to 48.1] | 0 [0.0 to 52.2] | 13 [1.7 to 40.5]
  IgG - Day 29 | 20 [4.3 to 48.1] | 53 [26.6 to 78.7] | 0 [0.0 to 52.2] | 0 [0.0 to 21.8]
  IgG - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgG - Day 181 | 17 [2.1 to 48.4] | 47 [21.3 to 73.4] | 0 [0.0 to 52.2] | 7 [0.2 to 33.9]
Statistical Analysis 1: Comparison: BPZE1 10^7 CFU by VaxINator vs Placebo by VaxINator; IgA, any time point; Test type: Superiority; p = 0.174, Barnard's exact test
Statistical Analysis 2: Comparison: BPZE1 10^9 CFU by VaxINator vs Placebo by VaxINator; IgA, any time point; Test type: Superiority; p = 0.006, Barnard's exact test
Statistical Analysis 3: Comparison: BPZE1 10^7 CFU by VaxINator vs Placebo by VaxINator; IgG, any time point; Test type: Superiority; p = 0.745, Barnard's exact test
Statistical Analysis 4: Comparison: BPZE1 10^9 CFU by VaxINator vs Placebo by VaxINator; IgG, any time point; Test type: Superiority; p = 0.023, Barnard's exact test

25. Secondary Outcome: Geometric Mean Titer Ratio of Mucosal FHA-IgA to Total IgA by Nasal Aspirate
Description: Nasal aspirate samples were collected from all participants at screening (baseline), Day 29, and Day 181 to measure total mucosal IgA levels via ELISA assay and mucosal IgA levels to filamentous hemagglutinin (FHA) pertussis antigen via a bead-based assay. Total mucosal IgA levels were reported in µg/mL; antigen-specific IgA results were reported in ELISA units/mL.
  The ratio of FHA-IgA to total mucosal IgA was computed for each participant and the geometric mean of the ratio was calculated for each study arm.
Time Frame: Screening, Day 29, Day 181
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titer Ratio
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
Titer Ratio
  Screening | 0.0154 [0.0104 to 0.0230] | 0.0133 [0.0098 to 0.0180] | 0.0251 [0.0025 to 0.2497] | 0.0147 [0.0093 to 0.0232]
  Day 29 | 0.0178 [0.0120 to 0.0264] | 0.0229 [0.0141 to 0.0372] | 0.0069 [0.0018 to 0.0271] | 0.0154 [0.0092 to 0.0258]
  Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  Day 181 | 0.011 [0.0062 to 0.0195] | 0.0263 [0.0155 to 0.0446] | 0.0109 [0.0038 to 0.0313] | 0.0185 [0.0102 to 0.0334]

26. Secondary Outcome: Geometric Mean Titer Ratio of Mucosal FIM-IgA to Total IgA by Nasal Aspirate
Description: Nasal aspirate samples were collected from all participants at screening (baseline), Day 29, and Day 181 to measure total mucosal IgA levels via ELISA assay and mucosal IgA levels to fimbriae 2/3 (FIM) pertussis antigen via a bead-based assay. Total mucosal IgA levels were reported in µg/mL; antigen-specific IgA results were reported in ELISA units/mL.
  The ratio of FIM-IgA to total mucosal IgA was computed for each participant and the geometric mean of the ratio was calculated for each study arm.
Time Frame: Screening, Day 29, Day 181
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titer Ratio
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
Titer Ratio
  Screening | 0.0023 [0.0010 to 0.0051] | 0.0012 [0.0005 to 0.0025] | 0.0073 [0.0005 to 0.1143] | 0.0023 [0.0010 to 0.0050]
  Day 29 | 0.0039 [0.0017 to 0.0090] | 0.0073 [0.0038 to 0.0139] | 0.0052 [0.0013 to 0.0216] | 0.0015 [0.0006 to 0.0037]
  Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  Day 181 | 0.0021 [0.0008 to 0.0057] | 0.0078 [0.0044 to 0.0139] | 0.0074 [0.0031 to 0.0180] | 0.0017 [0.0006 to 0.0047]

27. Secondary Outcome: Geometric Mean Titer Ratio of Mucosal PRN-IgA to Total IgA by Nasal Aspirate
Description: Nasal aspirate samples were collected from all participants at screening (baseline), Day 29, and Day 181 to measure total mucosal IgA levels via ELISA assay and mucosal IgA levels to pertactin (PRN) pertussis antigen via a bead-based assay. Total mucosal IgA levels were reported in µg/mL; antigen-specific IgA results were reported in ELISA units/mL.
  The ratio of PRN-IgA to total mucosal IgA was computed for each participant and the geometric mean of the ratio was calculated for each study arm.
Time Frame: Screening, Day 29, Day 181
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titer Ratio
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
Titer Ratio
  Screening | 0.0167 [0.0106 to 0.0263] | 0.007 [0.0043 to 0.0115] | 0.0063 [0.0030 to 0.0133] | 0.0106 [0.0052 to 0.0216]
  Day 29 | 0.0186 [0.0117 to 0.0295] | 0.0231 [0.0106 to 0.0500] | 0.0083 [0.0003 to 0.2520] | 0.0087 [0.0043 to 0.0175]
  Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  Day 181 | 0.0157 [0.0106 to 0.0233] | 0.0244 [0.0099 to 0.0602] | 0.0207 [0.0048 to 0.0892] | 0.0102 [0.0051 to 0.0204]

28. Secondary Outcome: Geometric Mean Titer Ratio of Mucosal PT-IgA to Total IgA by Nasal Aspirate
Description: Nasal aspirate samples were collected from all participants at screening (baseline), Day 29, and Day 181 to measure total mucosal IgA levels via ELISA assay and mucosal IgA levels to pertussis toxin (PT) pertussis antigen via a bead-based assay. Total mucosal IgA levels were reported in µg/mL; antigen-specific IgA results were reported in ELISA units/mL.
  The ratio of PT-IgA to total mucosal IgA was computed for each participant and the geometric mean of the ratio was calculated for each study arm.
Time Frame: Screening, Day 29, and Day 181
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titer Ratio
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
Titer Ratio
  Screening | 0.0014 [0.0009 to 0.0022] | 0.0011 [0.0007 to 0.0017] | 0.0021 [0.0015 to 0.0028] | 0.0011 [0.0007 to 0.0016]
  Day 29 | 0.0013 [0.0008 to 0.0020] | 0.0015 [0.0009 to 0.0026] | 0.0018 [0.0008 to 0.0039] | 0.0024 [0.0016 to 0.0036]
  Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  Day 181 | 0.0016 [0.0010 to 0.0024] | 0.0017 [0.0009 to 0.0031] | 0.0033 [0.0011 to 0.0098] | 0.0013 [0.0008 to 0.0024]

29. Secondary Outcome: Geometric Mean Titer by Serum IgA and Serum IgG to Filamentous Hemagglutinin
Description: Approximately 10 mL of venous blood was collected from participants immediately prior to the first study vaccination on Day 1 (baseline), Day 15, Day 29, and Day 181 to measure serum IgA and serum IgG levels (in ELISA units/mL) to filamentous hemagglutinin (FHA) pertussis antigen via a bead-based assay. The geometric mean FHA-IgA titer and FHA-IgG titer were calculated for each study arm.
Time Frame: Day 1, Day 15, Day 29, and Day 181
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
Titer
  IgA - Day 1 | 3.83 [1.40 to 10.48] | 3.54 [1.61 to 7.80] | 1.21 [0.25 to 5.95] | 2.71 [1.49 to 4.96]
  IgA - Day 15 | 3.06 [1.29 to 7.29] | 4.66 [2.12 to 10.24] | 1.75 [0.58 to 5.29] | 2.62 [1.50 to 4.55]
  IgA - Day 29 | 5.27 [2.46 to 11.29] | 8.67 [4.30 to 17.51] | 3.68 [1.20 to 11.28] | 2.21 [1.08 to 4.53]
  IgA - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgA - Day 181 | 5.13 [2.12 to 12.39] | 7.52 [3.57 to 15.85] | 2.81 [1.73 to 4.58] | 3.3 [1.66 to 6.57]
  IgG - Day 1 | 19.59 [8.04 to 47.69] | 19.65 [11.27 to 34.27] | 16.59 [2.33 to 118.01] | 12.81 [7.06 to 23.25]
  IgG - Day 15 | 19.99 [8.16 to 48.93] | 23.19 [16.00 to 33.62] | 12.78 [1.54 to 105.88] | 14.14 [7.10 to 28.14]
  IgG - Day 29 | 33.49 [16.56 to 67.72] | 29.4 [21.17 to 40.84] | 20.9 [2.90 to 150.52] | 11.96 [6.15 to 23.38]
  IgG - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgG - Day 181 | 32.73 [15.49 to 69.17] | 32.92 [24.18 to 44.83] | 19.62 [2.79 to 101.57] | 13.84 [6.22 to 30.80]

30. Secondary Outcome: Percentage of Participants Achieving Seroconversion to Pertactin as Measured by Serum IgA and Serum IgG Levels
Description: Approximately 10 mL of venous blood was collected from participants immediately prior to the first study vaccination on Day 1 (baseline), Day 15, Day 29, and Day 181 to measure via a bead-based assay serum IgA and serum IgG levels (in ELISA units/mL) to pertactin (PRN) pertussis antigen.
  Seroconversion was defined as at least a 2-fold rise in antigen-specific IgA and antigen-specific IgG levels post-baseline compared to baseline levels. The percentage of participants who seroconverted to PRN-IgA and PRN-IgG at any and each immunogenicity timepoint (Day 15, Day 29, or Day 181) were calculated.
Time Frame: Day 15, Day 29, and Day 181
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
percentage of participants
  IgA - Any Time Point | 13 [1.7 to 40.5] | 80 [51.9 to 95.7] | 40 [5.3 to 85.3] | 53 [26.6 to 78.7]
  IgA - Day 15 | 0 [0.0 to 21.8] | 40 [16.3 to 67.7] | 20 [0.5 to 71.6] | 13 [1.7 to 40.5]
  IgA - Day 29 | 13 [1.7 to 40.5] | 67 [38.4 to 88.2] | 40 [5.3 to 85.3] | 20 [4.3 to 48.1]
  IgA - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgA - Day 181 | 17 [2.1 to 48.4] | 67 [38.4 to 88.2] | 40 [5.3 to 85.3] | 36 [12.8 to 64.9]
  IgG - Any Time Point | 33 [11.8 to 61.6] | 47 [21.3 to 73.4] | 40 [5.3 to 85.3] | 20 [4.3 to 48.1]
  IgG - Day 15 | 7 [0.2 to 31.9] | 33 [11.8 to 61.6] | 0 [0.0 to 52.2] | 13 [1.7 to 40.5]
  IgG - Day 29 | 27 [7.8 to 55.1] | 40 [16.3 to 67.7] | 40 [5.3 to 85.3] | 7 [0.2 to 31.9]
  IgG - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgG - Day 181 | 25 [5.5 to 57.2] | 47 [21.3 to 73.4] | 0 [0.0 to 52.2] | 7 [0.2 to 33.9]
Statistical Analysis 1: Comparison: BPZE1 10^7 CFU by VaxINator vs Placebo by VaxINator; IgA, any time point; Test type: Superiority; p = 0.023, Barnard's exact test
Statistical Analysis 2: Comparison: BPZE1 10^9 CFU by VaxINator vs Placebo by VaxINator; IgA, any time point; Test type: Superiority; p = 0.142, Barnard's exact test
Statistical Analysis 3: Comparison: BPZE1 10^7 CFU by VaxINator vs Placebo by VaxINator; IgG, any time point; Test type: Superiority; p = 0.526, Barnard's exact test
Statistical Analysis 4: Comparison: BPZE1 10^9 CFU by VaxINator vs Placebo by VaxINator; IgG, any time point; Test type: Superiority; p = 0.142, Barnard's exact test

31. Secondary Outcome: Percentage of Participants Achieving Seroconversion to Pertussis Toxin as Measured by Serum IgA and Serum IgG Levels
Description: Approximately 10 mL of venous blood was collected from participants immediately prior to the first study vaccination on Day 1 (baseline), Day 15, Day 29, and Day 181 to measure via a bead-based assay serum IgA and serum IgG levels (in ELISA units/mL) to pertussis toxin (PT) antigen.
  Seroconversion was defined as at least a 2-fold rise in antigen-specific IgA/IgG levels post-baseline compared to baseline levels. The percentage of participants who seroconverted to PT-IgA and PT-IgG at any and each immunogenicity timepoint (Day 15, Day 29, or and Day 181) was calculated.
Time Frame: Day 15, Day 29, and Day 181
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
percentage of participants
  IgA - Any Time Point | 53 [26.6 to 78.7] | 60 [32.3 to 83.7] | 20 [0.5 to 71.6] | 60 [32.3 to 83.7]
  IgA - Day 15 | 13 [1.7 to 40.5] | 47 [21.3 to 73.4] | 20 [0.5 to 71.6] | 33 [11.8 to 61.6]
  IgA - Day 29 | 33 [11.8 to 61.6] | 47 [21.3 to 73.4] | 20 [0.5 to 71.6] | 33 [11.8 to 61.6]
  IgA - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgA - Day 181 | 17 [2.1 to 48.4] | 47 [21.3 to 73.4] | 20 [0.5 to 71.6] | 50 [23.0 to 77.0]
  IgG - Any Time Point | 27 [7.8 to 55.1] | 40 [16.3 to 67.7] | 20 [0.5 to 71.6] | 13 [1.7 to 40.5]
  IgG - Day 15 | 13 [1.7 to 40.5] | 13 [1.7 to 40.5] | 0 [0.0 to 52.2] | 7 [0.2 to 31.9]
  IgG - Day 29 | 13 [1.7 to 40.5] | 33 [11.8 to 61.6] | 20 [0.5 to 71.6] | 7 [0.2 to 31.9]
  IgG - Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  IgG - Day 181 | 25 [5.5 to 57.2] | 20 [4.3 to 48.1] | 20 [0.5 to 71.6] | 0 [0.0 to 23.2]
Statistical Analysis 1: Comparison: BPZE1 10^7 CFU by VaxINator vs Placebo by VaxINator; IgA, any time point; Test type: Superiority; p = 0.836, Barnard's exact test
Statistical Analysis 2: Comparison: BPZE1 10^9 CFU by VaxINator vs Placebo by VaxINator; IgA, any time point; Test type: Superiority; p = 1.000, Barnard's exact test
Statistical Analysis 3: Comparison: BPZE1 10^7 CFU by VaxINator vs Placebo by VaxINator; IgG, any time point; Test type: Superiority; p = 0.526, Barnard's exact test
Statistical Analysis 4: Comparison: BPZE1 10^9 CFU by VaxINator vs Placebo by VaxINator; IgG, any time point; Test type: Superiority; p = 0.119, Barnard's exact test

32. Secondary Outcome: Percentage of Participants Achieving Seroconversion to Filamentous Hemagglutinin as Measured by Mucosal IgA Levels
Description: Nasal aspirate samples were collected from all participants at screening (baseline), Day 29, and Day 181 to measure total mucosal IgA levels via ELISA assay and mucosal IgA levels to filamentous hemagglutinin (FHA) pertussis antigen via a bead-based assay. Total mucosal IgA levels were reported in µg/mL; antigen-specific IgA results were reported in ELISA units/mL.
  The titer ratio of antigen-specific IgA to total mucosal IgA was computed for each participant at each time point, and the fold rise from baseline of this ratio was subsequently calculated for each participant.
  Seroconversion was defined as at least a 2-fold rise in antigen-specific titer ratios post-baseline compared to baseline titer ratios. The percentage of participants who seroconverted FHA-IgA at each and any immunogenicity timepoint (Day 29 or Day 181) was calculated.
Time Frame: Day 29 and Day 181
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
percentage of participants
  Any Time Point | 20 [4.3 to 48.1] | 67 [38.4 to 88.2] | 40 [5.3 to 85.3] | 40 [16.3 to 67.7]
  Day 29 | 20 [4.3 to 48.1] | 47 [21.3 to 73.4] | 20 [0.5 to 71.6] | 7 [0.2 to 31.9]
  Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  Day 181 | 8 [0.2 to 38.5] | 53 [26.6 to 78.7] | 20 [0.5 to 71.6] | 43 [17.7 to 71.1]
Statistical Analysis 1: Comparison: BPZE1 10^7 CFU by VaxINator vs Placebo by VaxINator; Any time point; Test type: Superiority; p = 0.271, Barnard's exact test
Statistical Analysis 2: Comparison: BPZE1 10^9 CFU by VaxINator vs Placebo by VaxINator; Any time point; Test type: Superiority; p = 0.226, Barnard's exact test

33. Secondary Outcome: Percentage of Participants Achieving Seroconversion to Fimbriae 2/3 as Measured by Mucosal IgA Levels
Description: Nasal aspirate samples were collected from all participants at screening (baseline), Day 29, and Day 181 to measure total mucosal IgA levels via ELISA assay and mucosal IgA levels to fimbriae 2/3 (FIM) pertussis antigen via a bead-based assay. Total mucosal IgA levels were reported in µg/mL; antigen-specific IgA results were reported in ELISA units/mL.
  The titer ratio of antigen-specific IgA to total mucosal IgA was computed for each participant at each time point, and the fold rise from baseline of this ratio was subsequently calculated for each participant.
  Seroconversion was defined as at least a 2-fold rise in antigen-specific titer ratios post-baseline compared to baseline titer ratios. The percentage of participants who seroconverted FIM-IgA at each and any immunogenicity timepoint (Day 29 and Day 181) was calculated.
Time Frame: Day 29 and Day 181
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
percentage of participants
  Any Time Point | 27 [7.8 to 55.1] | 80 [51.9 to 95.7] | 60 [14.7 to 94.7] | 20 [4.3 to 48.1]
  Day 29 | 27 [7.8 to 55.1] | 53 [26.6 to 78.7] | 40 [5.3 to 85.3] | 7 [0.2 to 31.9]
  Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  Day 181 | 8 [0.2 to 38.5] | 80 [51.9 to 95.7] | 60 [14.7 to 94.7] | 14 [1.8 to 42.8]
Statistical Analysis 1: Comparison: BPZE1 10^7 CFU by VaxINator vs Placebo by VaxINator; Any time point; Test type: Superiority; p = 0.783, Barnard's exact test
Statistical Analysis 2: Comparison: BPZE1 10^9 CFU by VaxINator vs Placebo by VaxINator; Any time point; Test type: Superiority; p = 0.001, Barnard's exact test

34. Secondary Outcome: Percentage of Participants Achieving Seroconversion to Pertactin as Measured by Mucosal IgA Levels
Description: Nasal aspirate samples were collected from all participants at screening (baseline), Day 29, and Day 181 to measure total mucosal IgA levels via ELISA assay and mucosal IgA levels to pertactin (PRN) pertussis antigen via a bead-based assay. Total mucosal IgA levels were reported in µg/mL; antigen-specific IgA results were reported in ELISA units/mL.
  The titer ratio of antigen-specific IgA to total mucosal IgA was computed for each participant at each time point, and the fold rise from baseline of this ratio was subsequently calculated for each participant.
  Seroconversion was defined as at least a 2-fold rise in antigen-specific titer ratios post-baseline compared to baseline titer ratios. The percentage of participants who seroconverted PRN-IgA at each and any immunogenicity timepoint (Day 29 and Day 181) was calculated.
Time Frame: Day 29 and Day 181
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
percentage of participants
  Any Time Point | 13 [1.7 to 40.5] | 53 [26.6 to 78.7] | 80 [28.4 to 99.5] | 20 [4.3 to 48.1]
  Day 29 | 13 [1.7 to 40.5] | 40 [16.3 to 67.7] | 60 [14.7 to 94.7] | 13 [1.7 to 40.5]
  Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  Day 181 | 8 [0.2 to 38.5] | 47 [21.3 to 73.4] | 80 [28.4 to 99.5] | 21 [4.7 to 50.8]
Statistical Analysis 1: Comparison: BPZE1 10^7 CFU by VaxINator vs Placebo by VaxINator; Any time point; Test type: Superiority; p = 0.745, Barnard's exact test
Statistical Analysis 2: Comparison: BPZE1 10^9 CFU by VaxINator vs Placebo by VaxINator; Any time point; Test type: Superiority; p = 0.068, Barnard's exact test

35. Secondary Outcome: Percentage of Participants Achieving Seroconversion to Pertussis Toxin as Measured by Mucosal IgA Levels
Description: Nasal aspirate samples were collected from all participants at screening (baseline), Day 29, and Day 181 to measure total mucosal IgA levels via ELISA assay and mucosal IgA levels to pertussis toxin (PT) pertussis antigen via a bead-based assay. Total mucosal IgA levels were reported in µg/mL; antigen-specific IgA results were reported in ELISA units/mL.
  The titer ratio of antigen-specific IgA to total mucosal IgA was calculated for each participant at each time point, and the fold rise from baseline of this ratio was subsequently calculated for each participant.
  Seroconversion was defined as at least a 2-fold rise in antigen-specific titer ratios post-baseline compared to baseline titer ratios. The percentage of participants who seroconverted PT-IgA at each immunogenicity timepoint (Day 29 and Day 181) was calculated.
Time Frame: Day 29 and Day 181
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
percentage of participants
  Any Time Point | 40 [16.3 to 67.7] | 53 [26.6 to 78.7] | 20 [0.5 to 71.6] | 53 [26.6 to 78.7]
  Day 29 | 13 [1.7 to 40.5] | 33 [11.8 to 61.6] | 0 [0.0 to 52.2] | 53 [26.6 to 78.7]
  Day 181: number analyzed (Participants) | 12 | 15 | 5 | 14
  Day 181 | 42 [15.2 to 72.3] | 40 [16.3 to 67.7] | 20 [0.5 to 71.6] | 14 [1.8 to 42.8]
Statistical Analysis 1: Comparison: BPZE1 10^7 CFU by VaxINator vs Placebo by VaxINator; Any time point; Test type: Superiority; p = 0.585, Barnard's exact test
Statistical Analysis 2: Comparison: BPZE1 10^9 CFU by VaxINator vs Placebo by VaxINator; Any time point; Test type: Superiority; p = 1.000, Barnard's exact test

36. Primary Outcome: Number of Participants Experiencing Severe Solicited Systemic Reactogenicity AEs
Description: Solicited systemic reactogenicity events include fever, feverishness, fatigue, malaise, myalgia, arthralgia, headache, and rash/hypersensitivity. They were graded as grade 1 (mild), grade 2 (moderate), and grade 3 (severe). For all symptoms except rash and fever, an event was considered severe if it caused significant interference and prevented daily activity. Severe rash/hypersensitivity events were those that caused generalized urticaria, anaphylaxis, or angioedema or localized urticaria that required medical encounter. Severe fever was a temperature exceeding 38.9°C.
Time Frame: Day 1 through Day 15
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
Number analyzed (Participants) | 15 | 15 | 5 | 15
Participants
  Fever | 0 | 0 | 0 | 0
  Feverishness | 0 | 0 | 0 | 0
  Fatigue (tiredness) | 0 | 0 | 0 | 0
  Malaise (general unwell feeling) | 0 | 0 | 0 | 0
  Myalgia (body aches/muscular pain) | 0 | 0 | 0 | 0
  Arthralgia (joint pain) | 0 | 0 | 0 | 0
  Headache | 0 | 0 | 0 | 0
  Rash/hypersensitivity | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from the time of vaccination through approximately 6 months after vaccination. Solicited Adverse Events were collected from the time of each study vaccination through 14 days after study vaccination. Unsolicited AEs were collected from the time of study vaccination through approximately 28 days after study vaccination. New onset chronic medical conditions and adverse events of special interest were assessed through the follow-up period.
Description: Reactogenicity assessments included an assessment of solicited adverse events which includes an assessment of mucosal reactions that include: runny nose, stuffy nose/congestion, nasal pain/irritation, epistaxis, sneezing, sinus pressure/pain, sore throat, cough, and shortness of breath, as well as systemic reactions that include fever, chills, fatigue, malaise, myalgia, arthralgia, headache, and hypersensitivity.
Arm/Group | BPZE1 10^7 CFU by VaxINator | BPZE1 10^9 CFU by VaxINator | BPZE1 10^9 CFU by Syringe | Placebo by VaxINator
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/5 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/5 | 0/15
Other Adverse Events (participants affected / at risk) | 11/15 | 14/15 | 3/5 | 13/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BPZE1 10^7 CFU by VaxINator (N=15) | BPZE1 10^9 CFU by VaxINator (N=15) | BPZE1 10^9 CFU by Syringe (N=5) | Placebo by VaxINator (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (4) | 4 (4) | 2 (2) | 5 (5)
Feeling hot (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Malaise (General disorders) | 3 (3) | 3 (3) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Platelet count increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 9 (10) | 2 (2) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 8 (8) | 2 (2) | 6 (6)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 2 (2) | 3 (4)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 7 (7) | 2 (2) | 5 (6)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 1 (1) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT03541499/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/99/NCT03541499/SAP_001.pdf